CLINICAL TRIAL: NCT02801877
Title: Artificial Intelligence in a Mobile (AIM) Intervention for Depression
Brief Title: IntelliCare Study: Artificial Intelligence in a Mobile (AIM) Intervention for Depression
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH100482-01-RCTIC; R01MH100482-01 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety; Behavior Therapy; Technology Assisted; Mobile Phone; Cellular Phone; Smartphone; App; Coach
MeSH Terms: conditions — Depression; Anxiety Disorders; Alzheimer Disease | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IntelliCare Hub recommender, coach (Experimental): Participant is randomly assigned to receive the IntelliCare Hub App with the recommender system, and receive coaching for the 8 week IntelliCare program.
  Interventions: Behavioral: IntelliCare; Behavioral: Hub App with the Recommender System; Behavioral: Coaching
- IntelliCare Hub recommender, no coach (Experimental): Participant is randomly assigned to receive the IntelliCare Hub App with the recommender system, and independently use the IntelliCare program for 8 weeks.
  Interventions: Behavioral: IntelliCare; Behavioral: Hub App with the Recommender System
- IntelliCare Hub no recommender, coach (Experimental): Participant is randomly assigned to receive the IntelliCare Hub App without the recommender system, and receive coaching for the 8 week IntelliCare program.
  Interventions: Behavioral: IntelliCare; Behavioral: Coaching
- IntelliCare Hub no recommender, no coach (Experimental): Participant is randomly assigned to receive the IntelliCare Hub App without the recommender system, and independently use the IntelliCare program for 8 weeks.
  Interventions: Behavioral: IntelliCare

INTERVENTIONS:
Behavioral: IntelliCare
  Other Names: Behavioral intervention for depression & anxiety via app
Behavioral: Hub App with the Recommender System
  Other Names: Recommender via IntelliCare Hub app.
  Arms: IntelliCare Hub recommender, coach; IntelliCare Hub recommender, no coach
Behavioral: Coaching
  Other Names: Support from coach via phone calls and messaging
  Arms: IntelliCare Hub no recommender, coach; IntelliCare Hub recommender, coach

SUMMARY:
This study will evaluate and compare a smartphone intervention for depression and anxiety that uses machine learning to tailor treatment for participants with the same intervention without the machine learning component. The intervention, referred to as IntelliCare, delivers participant-specific treatment material and motivational messaging via a mobile phone to help individuals with depression and/or anxiety. Information and data received from the participant will inform the tailored treatment approach through machine learning. The purpose of this study is to compare different versions of the main IntelliCare Hub App (the centralized program delivery system) and participant user experience whether with the support of a coach or used independently. The randomized clinical trial (RCT) aims to obtain information on the feasibility and effectiveness of IntelliCare in improving symptoms of depression and anxiety.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common mental disorder, with up to 10.3% of the population experiencing the disorder in a given 12-month period. The relationship between depression and anxiety has been well documented. Depression is a significant predictor of future anxiety, and anxiety is a significant predictor of future onset of depression. Indeed, studies find that more than 50% of all individuals with MDD also have a current anxiety disorder. Although effective treatments have been developed over the years to address depression and anxiety, the lack of personalization and inability to adapt to patient needs or preferences contributes to poor treatment adherence and outcomes.

An intelligent treatment system was developed that uses state of the art machine learning approaches within a mobile intervention application to treat MDD and anxiety. Machine learning, a branch of artificial intelligence, focuses on the development of algorithms that automatically improve and evolve based on collected data. The intervention, called IntelliCare, uses a mobile application to continuously collect patient data and adapt intervention content and motivational messaging to create a highly tailored and user-responsive treatment system.

During the RCT study, 270 participants with Major Depression and/or Anxiety will use IntelliCare apps for up to 8 weeks and will be invited to complete online questionnaires at four follow-up time points: weeks 4 and 8 in the study program, and months 3 and 6 after the study program ends. All participants will first undergo initial assessments that will include a telephone interview and a series of online questionnaires about their mood. Eligible participants will receive up to 8 weeks of access to the IntelliCare system, which consists of apps with lessons and tools designed to teach skills for mood management. It is suggested that participants utilize the mobile phone tools every day.

Participants will be randomly assigned to one of two versions of the IntelliCare Hub App, which is the central delivery system for the IntelliCare program, and participants will also be randomly assigned to get support from a human coach or use the IntelliCare program independently.

Each week, participants assigned to work with a coach will receive a brief motivational intervention. This coach will also be available to participants via email throughout the 8 week study. Participants randomly assigned to use the IntelliCare program independently will receive an on-boarding guide to set up the IntelliCare Hub App on their phone, and participants will have access to our tech support team if technical difficulties arise while using the program.

Data from the RCT study will be used to examine whether: the IntelliCare program is an effective intervention for reducing depressive and anxiety symptoms; the recommender system will produce greater program adherence and; support from a coach or independent use might affect user experience and adherence. Data collected will also be used to further develop and evaluate machine learning methods for future research and deployment efforts.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for clinically significant symptoms of depression and/or anxiety using self-report measures used in screening for depression
* Is familiar with the use of mobile phones
* Owns an Android smartphone and is willing download the IntelliCare apps on their own device
* Is able to speak and read English
* Is at least 18 years of age (* Note: Depending on which state individual resides in, the age to consent to research may be 19 years of age.)
* Is able to give informed consent

Exclusion Criteria:

Participants were excluded if they had visual, voice, motor or hearing impairments that would prevent participation; met diagnostic criteria for a severe psychiatric disorders for which study treatments would be inappropriate; severe suicidality that included both a plan and intent; had initiated or modified antidepressant pharmacotherapy in the previous 14 days; or had used any IntelliCare app more than one time in the three months prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Interested parties may contact the PI. Data sharing may be considered if the proposed use is consistent with the protocol approved by the IRB and a Data Use Agreement is in place.

REFERENCES:
- [Derived] Mohr DC, Schueller SM, Tomasino KN, Kaiser SM, Alam N, Karr C, Vergara JL, Gray EL, Kwasny MJ, Lattie EG. Comparison of the Effects of Coaching and Receipt of App Recommendations on Depression, Anxiety, and Engagement in the IntelliCare Platform: Factorial Randomized Controlled Trial. J Med Internet Res. 2019 Aug 28;21(8):e13609. doi: 10.2196/13609. PMID 31464192

RESULTS

PARTICIPANT FLOW:
Groups:
- IntelliCare Hub Recommender, Coach: Participant is randomly assigned to receive the IntelliCare Hub App with the recommender system, and receive coaching for the 8 week IntelliCare program.
  IntelliCare
  Hub App with the Recommender System
  Coaching
- IntelliCare Hub Recommender, no Coach: Participant is randomly assigned to receive the IntelliCare Hub App with the recommender system, and independently use the IntelliCare program for 8 weeks.
  IntelliCare
  Hub App with the Recommender System
- IntelliCare Hub no Recommender, Coach: Participant is randomly assigned to receive the IntelliCare Hub App without the recommender system, and receive coaching for the 8 week IntelliCare program.
  IntelliCare
  Coaching
- IntelliCare Hub no Recommender, no Coach: Participant is randomly assigned to receive the IntelliCare Hub App without the recommender system, and independently use the IntelliCare program for 8 weeks.
  IntelliCare
Period: Overall Study
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach
Started | 74 | 75 | 76 | 76
Completed | 71 | 74 | 70 | 76
Not Completed | 3 | 1 | 6 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0
Not completed — Never Started Treatment | 2 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach | Total
Number analyzed (Participants) | 74 | 75 | 76 | 76 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (12.2) | 36.2 (11.5) | 37.1 (12.3) | 35.3 (11.5) | 36.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were provided option to not answer, or to answer not applicable.
  Participants
    number analyzed (Participants) | 72 | 75 | 76 | 76 | 299
    Female | 57 | 54 | 62 | 55 | 228
    Male | 15 | 21 | 14 | 21 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 7 | 5 | 30
  Not Hispanic or Latino | 62 | 67 | 68 | 71 | 268
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 5 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 8 | 6 | 29
  White | 57 | 63 | 57 | 60 | 237
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 6 | 8 | 25
Patient Health Questionaire 9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — A nine-item scale that assesses how often the respondent felt depressed over the last two weeks. Each item is scored on 0, not at all-3, nearly every day. The total score on the scale ranges from 0 (no depression) to 27 (severe depression).
  units on a scale | 12.78 (4.45) | 13.24 (4.55) | 13.11 (4.75) | 13.70 (4.79) | 13.21 (4.63)
Generalized Anxiety Disorder 7 (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — A 7 item scale that measures how often a respondent has felt anxious over the past 2 weeks. Each item is scored on a 0 (not at all)-3 (nearly every day) scale. The total score ranges from 0 (Not anxious) to 21 (Very anxious)
  units on a scale | 11.86 (4.05) | 11.88 (3.85) | 12.33 (4.51) | 11.84 (3.66) | 11.98 (4.02)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to the Mobile Application Intervention
Description: Defined as the median time to last engagement with the mobile application suite within 8 weeks of trial
Time Frame: Participants will be followed for the duration of the 8 week trial
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach
Number analyzed (Participants) | 74 | 75 | 76 | 76
days | 56 [56 to 56] | 56 [56 to 56] | 56 [55 to 56] | 56 [53 to 56]
Statistical Analysis 1: Comparison: IntelliCare Hub Recommender, Coach vs IntelliCare Hub Recommender, no Coach vs IntelliCare Hub no Recommender, Coach vs IntelliCare Hub no Recommender, no Coach; Log-rank test of adherence, defined as time to last engagement with mobile application suite; Test type: Superiority; p = 0.3, Log Rank; Chi square= 4.1 on 3 degrees of freedom

2. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9) - Depression Severity
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome. Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe.
Time Frame: Measured at start of treatment (baseline), week 4, week 8, month 3, and month 6.
Population: Participants with at least one follow-up measure of self-reported depression
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach
Number analyzed (Participants) | 71 | 74 | 70 | 76
score on a scale
  Week 4 | 8.87 (0.52) | 9.43 (0.51) | 8.82 (0.53) | 8.89 (0.51)
  Week 8 | 6.58 (0.52) | 7.90 (0.51) | 7.76 (0.53) | 8.20 (0.51)
  Month 3 (post treatment) | 6.52 (0.52) | 7.73 (0.51) | 7.62 (0.53) | 8.31 (0.51)
  Month 6 (post treatment) | 6.84 (0.53) | 8.35 (0.51) | 7.33 (0.53) | 7.72 (0.51)
Statistical Analysis 1: Comparison: IntelliCare Hub Recommender, Coach vs IntelliCare Hub Recommender, no Coach vs IntelliCare Hub no Recommender, Coach vs IntelliCare Hub no Recommender, no Coach; Interactive effect of time and group, adjusting for baseline PHQ-9, randomization strata, main and interactive effects of time, coach, coach*time, hub, and hub*time; Test type: Superiority; p = 0.90, Mixed Models Analysis; F(3, 835)=0.19

3. Primary Outcome: GAD-7 (Generalized Anxiety Disorder Scale-7) - Anxiety Severity
Description: The GAD-7 is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. GAD-7 total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome. Specifically, scores of 1-4 indicate minimal anxiety symptoms; 5-9 is mild anxiety symptoms; 10-14 is moderate anxiety symptoms; and 15-21 is severe anxiety symptoms.
Time Frame: Measured at start of treatment (baseline), week 4, week 8, month 3, and month 6.
Population: Participants with at least one follow-up measure of self-reported anxiety
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach
Number analyzed (Participants) | 71 | 74 | 70 | 76
score on a scale
  Week 4 | 7.66 (0.49) | 8.68 (0.48) | 7.67 (0.48) | 7.80 (0.48)
  Week 8 | 6.14 (0.49) | 7.68 (0.48) | 6.88 (0.48) | 7.04 (0.48)
  Month 3 (post treatment) | 5.70 (0.49) | 7.28 (0.48) | 6.45 (0.48) | 6.90 (0.49)
  Month 6 (post treatment) | 6.09 (0.49) | 6.99 (0.49) | 6.00 (0.48) | 6.83 (0.48)
Statistical Analysis 1: Comparison: IntelliCare Hub Recommender, Coach vs IntelliCare Hub Recommender, no Coach vs IntelliCare Hub no Recommender, Coach vs IntelliCare Hub no Recommender, no Coach; Interactive effect of time and group, adjusting for baseline GAD-7, randomization strata, main and interactive effects of time, coach, coach*time, hub, and hub*time; Test type: Superiority; p = 0.53, Mixed Models Analysis; F(3, 835)=0.73

ADVERSE EVENTS:
Time Frame: Screening through 6 months post treatment
Arm/Group | IntelliCare Hub Recommender, Coach | IntelliCare Hub Recommender, no Coach | IntelliCare Hub no Recommender, Coach | IntelliCare Hub no Recommender, no Coach
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/75 | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/74 | 0/75 | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT02801877/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02801877/ICF_001.pdf